CLINICAL TRIAL: NCT06960863
Title: Transient Elastography (Fibroscan) for Evaluation of Immunotherapy Response in Hepatocellular Carcinoma.
Brief Title: Fibroscan Evaluating Immunotherapy Response in Hepatocellular Carcinoma
Status: Recruiting | Type: Observational
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Rania Mamdouh Elkafoury, lecturer of Tropical medicine, Tanta University
Other Study IDs: 36264PR1126/3/25
Record Dates: First submitted 2025-04-29; First posted 2025-05-07 (Actual); Last update posted 2025-05-07 (Actual); Status verified 2025-04

CONDITIONS: Hepato Cellular Carcinoma (HCC)
Keywords: fibroscan; immunotherapy; liver stiffness; hepatocellular carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- HCC patients at baseline: At baseline, patients will undergo history-taking, clinical examination, laboratory investigations, Child-Pugh classification, Model for End-stage Liver Disease (MELD) score, BCLC staging, abdominal ultrasonography, Triphasic CT abdomen with contrast or MRI (for evaluation of tumor site, size and number), and Fibroscan examination
  Interventions: Radiation: fibroscan
- HCC patients 6 months post immunotherapy: All patients will be followed up after 6 months with clinic visits including laboratory testing, evaluation of treatment-related side effects, imaging studies, and fibroscan examination.
  Interventions: Radiation: fibroscan

INTERVENTIONS:
Radiation: fibroscan — Liver fibrosis and steatosis can be staged using Dimensional ultrasound TE (transient elastography).

SUMMARY:
The goal of this prospective cohort study is to evaluate the role of transient elastography (Fibroscan) in predicting the response of immunotherapy in advanced Hepatocellular carcinoma (HCC) patients.

Researchers will predict the response to 6 months of HCC immunotherapy regarding improvement of the degree of liver fibrosis, development of liver decompensation, complications, survival, and mortality.

Participants will undergo history-taking, clinical examination, laboratory investigations, Child-Pugh classification, Model for End-stage Liver Disease (MELD) score, BCLC staging, abdominal ultrasonography, Triphasic CT abdomen with contrast or MRI (for evaluation of tumor site, size and number), and Fibroscan examination at baseline and follow-up after 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients with confirmed advanced HCC (Diagnosed by two imaging modalities or liver biopsy) eligible for immunotherapy.
* Patients with preserved liver function (compensated Child-Pugh A if there is underlying cirrhosis).
* Patients with performance status ≤2 at staging work-up.
* absence of high-risk stigmata for bleeding on upper endoscopy, e.g. properly treated oesophageal varices and no history of variceal bleeding, in order to minimise bleeding risk.

Exclusion Criteria:

* Prior locoregional therapy or liver transplantation.
* Child-Pugh class C patients.
* Patients with performance status >2 at staging work-up.
* Vascular disorders, arterial hypertension, and risk of variceal bleeding.
* Severe autoimmune disorders.
* Patients who lost follow-up.
* Pregnant or breastfeeding women.
* Unwilling to participate in our study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This prospective cohort study will be carried out on 80 patients attending to Tanta tropical medicine outpatient clinic, faculty of medicine. The start of the research will be in January 2025 to January 2026 or until collecting the cases.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2025-01-26 (Actual); Primary Completion 2026-01-15 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Changes of liver stiffness measurement (kPa) | through study completion, an average of 1 year
  Measuring liver stiffness (kPa) using Fibroscan before and 6 months after immunotherapy.

SECONDARY OUTCOMES:
Decompensation rate | through study completion, an average of 1 year
  measuring liver decompensation rate after 6 months of immunotherapy
Mortality rate at 6 months follow-up | through study completion, an average of 1 year
  assessing mortality rate after 6 months of immunotherapy

CONTACTS AND LOCATIONS:
Overall Officials: Nabila A Elgazzar, MD, Principal Investigator — Tropical medicine and infectious diseases Department, Faculty of Medicine, Tanta University
Locations (1):
- Tanta University Hospitals, Tanta, Gharbyea, Egypt